CLINICAL TRIAL: NCT05491928
Title: Treatment of Metastatic Cancer in Terminally Diagnosed Patients
Status: Available | Type: Expanded Access
Sponsor: Matrix Biomed, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MBI-23-01
Record Dates: First submitted 2022-07-30; First posted 2022-08-08 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — tempol

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Tempol — Tempol will be given as an adjunct to chemotherapy.
  Other Names: MBM-0-1 MBM-02

SUMMARY:
The objective is to provide terminally diagnosed patients with a last line of treatment while improving overall quality of life. Tempol can be added to any chemotherapy regimen to potentially reduce side effects and overcome chemoresistance.

DETAILED DESCRIPTION:
The objective is to provide terminally diagnosed patients assigned to palliative care and palliative chemotherapy a last line treatment with Tempol. In vivo studies have shown Tempol to work synergistically with a number of chemotherapy agents increasing treatment response and reducing chemoresistance. Additionally, Tempol has been shown to provide protection to non-cancerous cells allowing for increased chemotherapy dosing by reducing side effects. Tempol inhibits HIF-1/VEGF among others in cancerous cells while upregulating GSH/NrF2 among others in non-cancerous cells.

ELIGIBILITY:
Inclusion Criteria:

* metastatic terminally diagnosed cancer

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- UCHealth University of Colorado Cancer Center - Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Background] Ravizza R, Cereda E, Monti E, Gariboldi MB. The piperidine nitroxide Tempol potentiates the cytotoxic effects of temozolomide in human glioblastoma cells. Int J Oncol. 2004 Dec;25(6):1817-22. PMID 15547722